# Evaluation of the Effect of Three Types of Rapid Maxillary Expanders (conventional, Hybrid and MSE)a randomized controlled trial

NCT05446714

Date : January 28, 2022



# Evaluation of the Effect of Three Types of Rapid Maxillary Expanders (conventional, Hybrid and MSE) a randomized controlled trial

# **CBCT Study**

# Protocol submitted in partial fulfilment of the requirements for Academic Promotion Degree in Orthodontics

By

#### Mohamed Abd El-Rahman Shendy

B.D.S (Al- Azhar University, Cairo, Boys) 2003G

M.D.Sc (Al- Azhar University, Cairo, Boys) 2013G

D.D.Sc (Al- Azhar University, Cairo, Boys) 2018G

Lecturer, Department of Orthodontics

Faculty of Dental Medicine

Al- Azhar University

Cairo (Boys)

#### **Contributors**

Dr. Mohamed Abd El-Rahman Shendy Dr Ahr

Dr Ahmed Mohamed Abouelnour

Lecturer, Department of Orthodontics

Lecturer, Department of Orthodontics

Faculty of Dental Medicine, Boys, Cairo

Faculty of Dental Medicine, Boys, Cairo

Al-Azhar University

Al-Azhar University

Department of Orthodontics

Faculty of Dental Medicine

Al- Azhar University

Cairo (Boys)

#### 2022G - 1443H

#### Introduction

Rapid maxillary expansion (RME)is a common procedure for correcting posterior crossbite, mild maxillary crowding and maxillary arch constriction through opening the mid palatal suture. (1-3)

RME can open the palatal and circum maxillary sutures, splitting of maxilla into two parts which affect nasal airway through increase nasal cavity volume followed by decreased nasal resistance and improved airflow especially in children with obstructive sleep apnea. (4-7)

Previous studies reported that RME can improve the airway (8-10)

On the other hand, other studies reported that RME does not affect oropharynx dimension. (11,12)

A systematic review mentioned that small changes in volume does not guaranty improvement in breathing mode, hence they advised the clinician not to do RME to improve the breathing mode. (13)

Current evidence suggested that the conflict might be the different protocols of CBCT between studies, Head posture, tongue position, and segmentation protocols were not standardized in the selected studies hence they recommended more accurate and reliable protocol with fixed head and tongue positioning, also the segmentation method. (14)

Other evidence showed improvement only limited to short term evaluation rather than long term one <sup>(15)</sup> While other evidence showed no improvement even with short term especially with miniscrew assisted rapid palatal expansion (MARPE). <sup>(16)</sup>

So the aim of this study was to evaluate the effect of three types of rapid maxillary expanders (conventional, Hybrid and MSE) using cone beam computed tomography (CBCT)

# Aim of study

The aim of this study was to compare the effect of three types of rapid maxillary expanders (conventional, Hybrid and MSE) using cone beam computed tomography (CBCT)

# The secondary outcomes

- a- Evaluation of periodontal condition of maxillary first permanent molars, both clinically and radiographically using CBCT
- b- Evaluation of Airway.

#### **Material and Methods**

# Study design:

Prospective randomized controlled trial

### Study setting and population:

This study will be conducted on patients seeking orthodontic treatment in the outpatient clinic, Orthodontic department, Faculty of Dental Medicine, Al-Azhar University, Cairo, Boys branch.

# Eligibility criteria of population:

The patients will be selected according to the following inclusions criteria:

- 1- Patients suffering maxillary collapse with a skeletal background
- 2- Patients with unilateral or bilateral posterior crossbite.
- 3- Patients with reduced or average anterior face height.
- 4- Patients with no periodontal disease.
- 5- Patients with good oral hygiene and general health.
- 6- No systemic diseases that may affect bone quality or interfere with orthodontic treatment.
- 7- Patients with erupted maxillary permanent first molars and premolars.
- 8- Patients with no previous orthodontic treatment.

# Sample size:

Sample size calculation using G power software was based on the observed effect sizes derived from previous article. (20)

The calculation indicated that for a study with a power of 0.95 and an alpha of 0.05, a total of at least 45 patients (15 patients in each group).

#### Group allocation:

The patients will be classified and randomly allocated into three equal groups, using online generated randomization plan (Graph Pad) found at the website

http://www.graphpad.com/quickcalcs/index.cfm.:

- Group (1): The conventional hyrax.
- Group (2): The Hybrid hyrax.
- Group (3): The MSE expander.

#### Interventions:

The current study was conducted on a total sample of forty five young adult orthodontic patients presented with transverse maxillary deficiency with an age ranged from 11-16 years.

- All patients in this study will undergo a special protocol for oral hygiene measures for one month to standardize as possible the oral hygiene measure before expansion.
- The following diagnostic records will be taken for each patient before and after the completion of expansion treatment:
- Orthodontic study casts.
- Standardized extra-oral and intra-oral photographs.
- Panoramic and Upper occlusal radiographs.
- Other radiographic evaluations that serve the purpose of the study according to the situation.

- Radiographic analysis will be performed for each patient to evaluate the effect of the rapid maxillary expansion on the nasal airway.

#### Ethical consideration:

The objectives of the study will be discussed to the patients and parents and informed consent will be signed before treatment (form is attached).

#### Data management and analysis:

- The collected data will be statistically analyzed using SPSS.

The Institutional Ethical Committee: approval number 775/220

#### References

- 1. Lagravere MO, Major PW, Flores-Mir C. Long-term skeletal changes with rapid maxillary expansion: a systematic review. Angle Orthod. 2005;75:1046–1052.-
- 2. Gracco A, Malaguti A, Lombardo L, Mazzoli A, Raffaelie R. Palatal volume following rapid maxillary expansion in mixed dentition. Angle Orthod.2010;80:153–9.
- 3. Jia H, Zhuang L, Zhang N, Bian Y, Li S. Age-dependent effects of transverse maxillary deficiency treated by microimplant-assisted rapid palatal expansion: A prospective cone-beam computed tomography study. Am J Orthod Dentofacial Orthop. 2021 Dec 10:S0889-5406(21)00730-7. doi: 10.1016/j.ajodo.2020.10.029. Epub ahead of print. PMID: 34903419.
- 4. Haas AJ. Rapid expansion of the maxillary dental arch and nasal cavity by opening the midpalatal suture. Angle Orthod. 1961;31(2):73-90.
- 5. Bazargani F, Feldmann I, Bondemark L. Three-dimensional analysis of effects of rapid maxillary expansion on facial sutures and bones: a systematic review. Angle Orthod. 2013;7(6):1074-82.

- 6. Mehta S, Wang D, Kuo CL, et al. Long-term effects of mini-screw-assisted rapid palatal expansion on airway. AngleOrthod. 2021;91:195–205.
- 7. Villa MP, Castaldo R, Miano S, Paolino MC, Vitelli O, Tabarrini A, Mazzotta AR, Cecili M, Barreto M. Adenotonsillectomy and orthodontic therapy in pediatric obstructive sleep apnea. Sleep Breath. 2014 Sep;18(3):533-9. doi: 10.1007/s11325-013-0915-3. Epub 2013 Nov 26. PMID: 24277354.
- 8. Buck LM, Dalci O, Darendeliler MA, Papageorgiou SN, Papadopoulou AK. Volumetric upper airway changes after rapid maxillary expansion: a systematic review and meta-analysis. European journal of orthodontics. 2017 Oct 1;39(5):463-73.
- 9. Bazargani F, Magnuson A, Ludwig B. Effects on nasal airflow and resistance using two different RME appliances: a randomized controlled trial. European Journal of Orthodontics. 2018 May 25;40(3):281-4.
- 10.Kavand G, Lagravère M, Kula K, Stewart K, Ghoneima A. Retrospective CBCT analysis of airway volume changes after boneborne vs tooth-borne rapid maxillary expansion. The Angle Orthodontist. 2019 Jul;89(4):566-74.
- 11. Abdalla Y, Brown L, Sonnesen L. Effects of rapid maxillary expansion on upper airway volume: A three-dimensional cone-beam computed tomography study. Angle Orthod. 2019 Nov;89(6):917-923. doi: 10.2319/101218-738.1. Epub 2019 Apr 3. PMID: 30942607; PMCID: PMC8109167.
- 12.El H, Palomo JM. Three-dimensional evaluation of upper airway following rapid maxillary expansion: a CBCT study. Angle Orthod. 2014 Mar;84(2):265-73. doi: 10.2319/012313-71.1. Epub 2013 Jul 18. PMID: 23865825; PMCID: PMC8673812.
- 13.Gordon JM, Rosenblatt M, Witmans M, Carey JP, Heo G, Major PW, Flores-Mir C. Rapid palatal expansion effects on nasal airway dimensions as measured by acoustic rhinometry: a systematic review. The Angle Orthodontist. 2009 Sep;79(5):1000-7.
- 14.Di Carlo G, Saccucci M, Ierardo G, Luzzi V, Occasi F, Zicari AM, Duse M, Polimeni A. Rapid maxillary expansion and upper airway morphology: a systematic review on the role of cone beam computed tomography. BioMed research international. 2017 Jul 16;2017.

- 15.Niu X, Di Carlo G, Cornelis MA, Cattaneo PM. Three-dimensional analyses of short-and long-term effects of rapid maxillary expansion on nasal cavity and upper airway: a systematic review and meta-analysis. Orthodontics & craniofacial research. 2020 Aug;23(3):250-76.
- 16.Arqub SA, Mehta S, Iverson MG, Yadav S, Upadhyay M, Almuzian M. Does Mini Screw Assisted Rapid Palatal Expansion (MARPE) have an influence on airway and breathing in middle-aged children and adolescents? A systematic review. International orthodontics. 2021 Mar 1;19(1):37-50.
- 17.Iwasaki T, Saitoh I, Takemoto Y, Inada E, Kakuno E, Kanomi R, Hayasaki H, Yamasaki Y. Tongue posture improvement and pharyngeal airway enlargement as secondary effects of rapid maxillary expansion: a cone-beam computed tomography study. Am J Orthod Dentofacial Orthop. 2013 Feb;143(2):235-45. doi: 10.1016/j.ajodo.2012.09.014. PMID: 23374931.
- 18.Baka ZM, Akin M, Ucar FI, Ileri Z. Cone-beam computed tomography evaluation of dentoskeletal changes after asymmetric rapid maxillary expansion. Am J Orthod Dentofacial Orthop. 2015 Jan;147(1):61-71. doi: 10.1016/j.ajodo.2014.09.014. PMID: 25533073.
- 19.Li Q, Tang H, Liu X, Luo Q, Jiang Z, Martin D, Guo J. Comparison of dimensions and volume of upper airway before and after minimplant assisted rapid maxillary expansion. Angle Orthod. 2020 May 1;90(3):432-441. doi: 10.2319/080919-522.1. PMID: 33378437; PMCID: PMC8032299.
- 20.Brunetto M, Andriani J da SP, Ribeiro GLU, Locks A, Correa M, Correa LR. Three-dimensional assessment of buccal alveolar bone after rapid and slow maxillary expansion: a clinical trial study. American Journal of Orthodontics and Dentofacial Orthopedics 2013;143(5):633–44.